CLINICAL TRIAL: NCT05533359
Title: SCALE-UP Utah II: Community-Academic Partnership to Address COVID-19 Testing and Vaccination Among Utah Community Health Centers
Brief Title: SCALE-UP Utah II: Community-Academic Partnership to Address COVID-19 Conversational Agent Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Utah Department of Health (Other); Association for Utah Community Health (Other); National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Guilherme Del Fiol, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 00150669_2; U01MD017421 (NIH)
Record Dates: First submitted 2022-09-07; First posted 2022-09-09 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Patient-level, four-arm randomized design for Population Health Management interventions: (1) TM + No PN, (2) TM + Request PN, (3) CA + No PN, or (4) CA + Request PN
Who Masked: Participant
Masking Description: Patients will not know what intervention arm they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Text Messaging (TM) + No Patient Navigation (Active Comparator): Bidirectional text messaging with a one-touch response to connect patients to vaccination or mailed at-home rapid test kits for use as needed.
  Patients will not receive patient navigation.
  Interventions: Behavioral: Text-Messaging (TM)
- Text Message (TM) + Request (RPN) (Active Comparator): Bidirectional text messaging with a one-touch response to connect patients to vaccination or mailed at-home rapid test kits for use as needed.
  RPN will provide patients the opportunity to reply PERSON (for connection to a PN) in response to a TM offering connection to testing and/or vaccination.
  Interventions: Behavioral: Text-Messaging (TM); Behavioral: Patient Navigation (PN)
- Conversational Agent (CA)+ No Patient Navigation (Active Comparator): Automated, scripted and interactive conversational agent used to mimic human interaction to: 1) elicit specific hesitancy factors and barriers to testing; 2) provide tailored information to address each individual's hesitancy factors and barriers to testing; and 3) offer access to at-home rapid test kits.
  Patients will not receive patient navigation.
  Interventions: Behavioral: Conversational Agent (CA)
- Conversational Agent (CA) + Request PN (RPN) (Active Comparator): Automated, scripted and interactive conversational agent used to mimic human interaction to: 1) elicit specific hesitancy factors and barriers to testing; 2) provide tailored information to address each individual's hesitancy factors and barriers to testing; and 3) offer access to at-home rapid test kits.
  RPN will provide patients the opportunity to reply PERSON (for connection to a PN) in response to a CA offering connection to testing and/or vaccination.
  Interventions: Behavioral: Conversational Agent (CA); Behavioral: Patient Navigation (PN)

INTERVENTIONS:
Behavioral: Text-Messaging (TM) — Participants in the TM condition will receive HIPAA-compliant bidirectional text messages. These texts will include a brief message alerting patients that they are eligible to receive a test kit and asking participants if they would like to receive a test kit. Participants who reply "yes" will receive an additional message with information about how to receive a test kit.
  Arms: Text Message (TM) + Request (RPN); Text Messaging (TM) + No Patient Navigation
Behavioral: Conversational Agent (CA) — Patients in the CA condition will receive a link to an automated, scripted and interactive conversational agent used to mimic human interaction to: 1) elicit specific hesitancy factors and barriers to testing; 2) provide tailored information to address each individual's hesitancy factors and barriers to testing; and 3) offer access to at-home rapid test kits.
  Arms: Conversational Agent (CA) + Request PN (RPN); Conversational Agent (CA)+ No Patient Navigation
Behavioral: Patient Navigation (PN) — Participants in the PN condition will receive a call from a Community Health Worker to assist with the process of receiving a COVID test. At this time the participant has the option to opt-out of this follow up phone call. The patient navigation from the Community Health Worker includes practical advice in addressing barriers to testing such as logistics, as well as fear, skepticism, and hesitancy.
  There are two distinct different types of patient navigation. A person can be randomly assigned to either type, or no PN, or a combination of the two types.
  Arms: Conversational Agent (CA) + Request PN (RPN); Text Message (TM) + Request (RPN)

SUMMARY:
The long-term objective of SCALE-UP II is to increase the reach, uptake, and sustainability of COVID-19 testing among underserved populations. Through RADx-UP Phase I funding (SCALE-UP Utah), the team has established population health management (PHM) interventions that have been used since Feb 2021 to increase the uptake of COVID-19 testing and vaccination among community health center patients.

Interventions are based on a PHM approach that uses widely available technology (i.e. cell phones and text messaging). SCALE-UP II will both build on SCALE-UP Utah PHM interventions and investigate novel resource conservation approaches (i.e., Request-Patient Navigation vs. No Patient Navigation and text messaging vs. conversational agent).

SCALE-UP II builds on long standing partnerships among the University of Utah Clinical and Translational Science Institute (UofU CTSI), Association for Utah Community Health (AUCH), CHCs, and the Utah Department of Health(UDOH). CTSI and SCALE-UP II investigators are leading several COVID-19 initiatives that drive public health response and state government policies in Utah. Thus, the UofU team is uniquely positioned to lead this project.

DETAILED DESCRIPTION:
Racial/ethnic minority, low socioeconomic status (SES), and rural populations suffer profound health inequities across a wide variety of diseases and conditions, including COVID-19. For example, as of June 2021, the cumulative COVID case rate in Utah per 100,000 was 10,803 among Whites vs. 17,541 among Latinos. The positivity rate was 14% among Whites vs. 24% among Latinos. Similar disparities persist across the nation for vaccination rates between urban vs. rural, high vs. low SES, and White vs. non-White populations. Low vaccination rates leave underserved populations at risk for local outbreaks, and more contagious and severe variants. Thus, interventions targeting these populations at the interplay between testing and vaccination among underserved populations are critical for pandemic control.

Not only do underserved populations experience profound health inequities, but there is also a critical digital divide between high and low resource healthcare systems. Low resource settings are far less likely to adopt Health Information Technology approaches, and often do not have the capacity to implement large scale population health management (PHM) efforts utilizing data analytics and automated patient outreach. As such, research is needed utilizing targeted PHM approaches that proactively identify, reach, and navigate vulnerable patients to both increase opportunities to engage in vaccination and testing, and to address barriers to engagement. Community Health Centers (CHCs) are optimal settings for implementation of PHM interventions to increase the uptake of COVID-19 testing and vaccination among underserved populations. Eleven Utah CHC systems are participating in SCALE-UP II. Their 38 primary care clinics serve over 112,000 unique patients annually (36% Latino, 10% Native American, 63% <100% poverty level, 57% uninsured, and 42% of clinics are in rural/frontier areas).

SCALE UP II is comprised of two distinct studies, the Text Message (TM) study and the Conversational Agent (CA) study. Patients will be triaged into one of two studies based on self-reported ownership of a smart phone with internet access. Patients who report not owning a smart phone with internet access will be included in the TM study. Additionally, patients who do not respond to the question regarding smart phone ownership will be included in the TM study. Patients who self-report ownership of a smart phone with internet access will be included in the CA study.

SCALE-UP II: CA study will implement and evaluate practical, accessible, and scalable PHM interventions to increase COVID-19 testing and vaccine uptake based on the best evidence available, patients' specific barriers and hesitancy factors, and extensive collaboration with CHCs, AUCH, and UDHHS. This study is a 2x2 design with patients being initially randomized between receiving either text messages or the link to a conversational agent as well as into two distinct types of available patient navigation, Request-PN or No PN.

Text Messaging (TM): bidirectional text messaging to connect patients to vaccination or mailed at-home rapid test kits for use, as needed.

Conversational Agent (CA): automated, scripted and interactive agent used to mimic human interaction to: 1) elicit specific hesitancy factors and barriers to testing; 2) provide tailored information to address each individual's hesitancy factors and barriers to testing; and 3) offer access to at-home rapid test kits.

Patient Navigation (PN): phone call from a community health worker to help address hesitancy and barriers, and to offer at-home rapid test kits. This study will examine two distinct forms of Patient Navigation: Request PN and No PN. Each patient will be randomized to receive either Request PN or No PN. Request PN allows patients to request patient navigation by responding PERSON to a text message/conversational agent. Patients who are randomized to receive No PN will not be provided the opportunity to speak with a patient navigator.

The primary outcome, Reach-Accept Testing, captures whether patients requests an at-home test kit and confirmed their mailing address. Secondary outcomes include: Testing (i.e. the proportion of participants who self-report having used an at-home test at least once during follow-up) as well as several implementation outcomes including Reach-Engage Testing (proportion of patients that reply to an offer to receive an at-home rapid test kit), PN-Request (proportion in PN who requested patient navigation), PN-Engage (proportion in PB who talked to a patient navigator), and Opt-Out. The outcomes and compared groups provided for the Smartphone study are main effects for delivery mechanism (Chatbot & TM), main effects for PN (PN & No PN), and main effects for message frequency (10-day & 30-day).

SCALE-UP II will include a Consortium Data Reporting Unit (CDRU) consisting of a Data Manager and one member the project's biomedical informatics team. The unit will attend regular meetings and dissemination activities organized by the CDCC. The CDRU will seek guidance from the CDCC with regard to data acquisition and consent for data sharing. As required by the NIH, SCALE-UP II will collect RADx-UP Tier 1 Common Data Elements for study participants who receive an at-home COVID test through the project. These data will be collected through surveys administered one month after the participant receives their at-home test. Data will be standardized according to the data dictionary provided by the CDCC. Our CDRU will work closely with the CDCC to establish a protocol for frequency, format, and exchange of data. SCALE-UP II will share identifiable data with the CDCC and NIH for the Data Hub as well as future research. Participants who complete the survey data will first complete an informed consent process. The informed consent will be administered to the patient at the time of survey collection.

Lighthouse Research and Development will conduct phone surveys to assess patient reported use of COVID-19 at-home testing (~2,300 participants) among patients who received test kits and do no respond to the online survey request. Lighthouse will send notifications (e.g., postcards, text messages, voice messages, etc.) to participants to alert them of the opportunity to complete the survey online or over the phone. Interviewers will complete up to 15 call attempts across weekday, evening, and weekend calling shifts over a one-month period to each participant. Patients will be compensated with a gift card for completing the survey.

ELIGIBILITY:
Inclusion Criteria:

* current patient of a participating community health center
* have a working cellphone,
* have phone number listed in existing electronic medical record at their participating clinic
* speak English or Spanish.

Exclusion Criteria:

* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2117 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Del Fiol, MD PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Fiol G, Kuzmenko TV, Orleans B, Chipman JJ, Greene T, Meads R, Kaphingst KA, Gibson B, Kawamoto K, King AJ, Siaperas T, Hughes S, Pruhs A, Dinkins CP, Lam CY, Pierce JH, Benson R, Borsato EP, Cornia RC, Stevens L, Bradshaw RL, Schlechter CR, Wetter DW. Population-Based Digital Health Interventions to Deliver at-Home COVID-19 Testing: SCALE-UP II Randomized Clinical Trial. J Med Internet Res. 2025 Jul 28;27:e74145. doi: 10.2196/74145. PMID 40720824
- [Derived] Del Fiol G, Orleans B, Kuzmenko TV, Chipman J, Greene T, Martinez A, Wirth J, Meads R, Kaphingst KK, Gibson B, Kawamoto K, King AJ, Siaperas T, Hughes S, Pruhs A, Pariera Dinkins C, Lam CY, Pierce JH, Benson R, Borsato EP, Cornia R, Stevens L, Bradshaw RL, Schlechter CR, Wetter DW. SCALE-UP II: protocol for a pragmatic randomised trial examining population health management interventions to increase the uptake of at-home COVID-19 testing in community health centres. BMJ Open. 2024 Mar 20;14(3):e081455. doi: 10.1136/bmjopen-2023-081455. PMID 38508633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited participants in partnership with the Association for Utah Community Health and its affiliated Community Health Centers (CHCs). Three CHCs with 12 primary care clinics participated. Eligible patients had an appointment at one of the participating CHCs in the last 3 years, were 18 years and older, and had a valid cellphone number in the CHC EHR. Specific to the Conversational Agent group: these patients had also replied to a TM that they did have a Smart Phone.
Pre-assignment Details: 1. Opted Out- opted out after receiving introductory text but before randomization
  2. Smart Phone- Participant responded that they do have a Smart Phone
Groups:
- Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day: Patients in this group received a link to an automated scripted and interactive conversation agent used to mimic human interaction to: 1) elicit specific hesitancy factors and barriers to testing; 2) provide tailored information to address each individual's hesitancy factors and barriers to testing; and 3) offer access to at-home rapid test kits. Participants in this group did not receive Patient Navigation, and outreach frequency was intervention message delivered every 10 days for a total of 6 messages.
- Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day: Patients in this group received a link to an automated scripted and interactive conversation agent used to mimic human interaction to: 1) elicit specific hesitancy factors and barriers to testing; 2) provide tailored information to address each individual's hesitancy factors and barriers to testing; and 3) offer access to at-home rapid test kits. Participants in this group did not receive Patient Navigation, and outreach frequency was intervention message delivered every 30 days for a total of 3 messages.
- Conversational Agent (CA) + Patient Navigation (PN) + 10 Day: Patients in this group received a link to an automated scripted and interactive conversation agent used to mimic human interaction to: 1) elicit specific hesitancy factors and barriers to testing; 2) provide tailored information to address each individual's hesitancy factors and barriers to testing; and 3) offer access to at-home rapid test kits. Participants in this group could receive Patient Navigation. Patient navigation was a phone call from a community health worker that gave practical advice in addressing barriers to testing. Outreach frequency was intervention message delivered every 10 days for a total of 6 messages.
- Conversational Agent (CA) + Patient Navigation (PN) + 30 Day: Patients in this group received a link to an automated scripted and interactive conversation agent used to mimic human interaction to: 1) elicit specific hesitancy factors and barriers to testing; 2) provide tailored information to address each individual's hesitancy factors and barriers to testing; and 3) offer access to at-home rapid test kits. Participants in this group could receive Patient Navigation. Patient navigation was a phone call from a community health worker that gave practical advice in addressing barriers to testing. Outreach frequency was intervention message delivered every 30 days for a total of 3 messages.
- Text Message (TM) + No Patient Navigation (NoPN) + 10 Day: Patients in this group received a bidirectional text message that included a brief message alerting patients they were eligible to receive a test kit. Participants in this group did not receive Patient Navigation, and outreach frequency was intervention message delivered every 10 days for a total of 6 messages.
- Text Message (TM) + No Patient Navigation (NoPN) + 30 Day: Patients in this group received a bidirectional text message that included a brief message alerting patients they were eligible to receive a test kit. Participants in this group did not receive Patient Navigation, and outreach frequency was intervention message delivered every 30 days for a total of 3 messages.
- Text Message (TM) + Patient Navigation (PN) + 10 Day: Patients in this group received a bidirectional text message that included a brief message alerting patients they were eligible to receive a test kit. Participants in this group could receive Patient Navigation. Patient navigation was a phone call from a community health worker that gave practical advice in addressing barriers to testing. Outreach frequency was intervention message delivered every 10 days for a total of 6 messages.
- Text Message (TM) + Patient Navigation (PN) + 30 Day: Patients in this group received a bidirectional text message that included a brief message alerting patients they were eligible to receive a test kit. Participants in this group could receive Patient Navigation. Patient navigation was a phone call from a community health worker that gave practical advice in addressing barriers to testing. Outreach frequency was intervention message delivered every 30 days for a total of 3 messages.
Period: Overall Study
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day
Started | 261 | 264 | 264 | 262 | 265 | 265 | 270 | 266
Completed | 247 | 262 | 237 | 249 | 242 | 262 | 255 | 257
Not Completed | 14 | 2 | 27 | 13 | 23 | 3 | 15 | 9

BASELINE CHARACTERISTICS:
Population: Analysis population are patients who had an appointment at one of the participating CHCs in the last three years, were 18 years and older, had a valid cellphone number recorded in the CHC electronic health record and had a Smart Phone.
Groups:
- Total: Total of all reporting groups
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day | Total
Number analyzed (Participants) | 261 | 264 | 264 | 262 | 265 | 265 | 270 | 266 | 2117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.38 (14.55) | 49.88 (15.38) | 48.83 (14.93) | 48.34 (14.23) | 48.89 (14.22) | 47.92 (14.40) | 49.79 (15.36) | 49.13 (13.85) | 49.02 (14.62)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 179 | 163 | 188 | 181 | 182 | 191 | 186 | 181 | 1451
  Sex: Male | 82 | 101 | 75 | 81 | 83 | 74 | 84 | 85 | 665
  Sex: Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ehtnicity: American Indian/Alaska Native | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
  Race/Ehtnicity: Asian | 1 | 1 | 3 | 0 | 1 | 3 | 1 | 4 | 14
  Race/Ehtnicity: Black/African American | 3 | 3 | 1 | 3 | 1 | 3 | 5 | 0 | 19
  Race/Ehtnicity: Hawaiian/Pacific Islander | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 8
  Race/Ehtnicity: Hispanic or Latino/a | 152 | 144 | 137 | 139 | 140 | 142 | 144 | 160 | 1158
  Race/Ehtnicity: Unknown | 19 | 22 | 25 | 21 | 21 | 22 | 22 | 19 | 171
  Race/Ehtnicity: White Non-Hispanic | 84 | 86 | 93 | 92 | 97 | 93 | 93 | 81 | 719
  Race/Ehtnicity: Multi-race | 1 | 6 | 4 | 5 | 3 | 2 | 4 | 0 | 25
Language [Count of Participants; unit: Participants]
  English | 125 | 128 | 127 | 141 | 124 | 134 | 130 | 117 | 1026
  Spanish | 123 | 126 | 123 | 113 | 128 | 121 | 125 | 134 | 993
  Other | 5 | 3 | 5 | 3 | 3 | 4 | 7 | 5 | 35
  Unknown | 8 | 7 | 9 | 5 | 10 | 6 | 8 | 10 | 63
Urban/Rural [Count of Participants; unit: Participants]
  Urban | 227 | 230 | 231 | 230 | 228 | 231 | 233 | 230 | 1840
  Rural | 34 | 34 | 33 | 32 | 37 | 34 | 37 | 36 | 277
Insurance Status [Count of Participants; unit: Participants]
  Private | 63 | 80 | 69 | 88 | 71 | 85 | 76 | 78 | 610
  Public | 47 | 44 | 44 | 45 | 43 | 38 | 40 | 42 | 343
  Uninsured | 151 | 140 | 151 | 129 | 151 | 142 | 154 | 146 | 1164
CHC [Count of Participants; unit: Participants] — Number of participating patients by CHC
  Participants
    CHC 1 | 160 | 162 | 165 | 162 | 163 | 162 | 166 | 166 | 1306
    CHC 2 | 35 | 36 | 34 | 33 | 36 | 34 | 36 | 34 | 278
    CHC 3 | 66 | 66 | 65 | 67 | 66 | 69 | 68 | 66 | 533
SCALE-UP I Randomization [Count of Participants; unit: Participants]
  Not enrolled in SCALE UP I | 83 | 81 | 82 | 80 | 86 | 83 | 86 | 83 | 664
  TM | 79 | 81 | 81 | 79 | 79 | 80 | 81 | 81 | 641
  TM+PN | 99 | 102 | 101 | 103 | 100 | 102 | 103 | 102 | 812

OUTCOME MEASURES:

1. Primary Outcome: Reach-Accept Testing
Description: Number of patients who requested a test kit and confirmed their mailing address.
Time Frame: Every 10 or 30 days dependent on group randomization [up to 90 days post intervention message] Every 10 or 30 days from intervention messaging for 90 days dependent on group randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day
Number analyzed (Participants) | 261 | 264 | 264 | 262 | 265 | 265 | 270 | 266
Participants | 47 | 41 | 41 | 45 | 142 | 139 | 151 | 123

2. Secondary Outcome: Reach-Engage Testing
Description: Number of patients that reply to an offer to receive an at-home rapid test kit
Time Frame: Every 10 or 30 days dependent on group randomization [up to 90 days post intervention message]
Measure: Count of Participants; unit: Participants
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day
Number analyzed (Participants) | 261 | 264 | 264 | 262 | 265 | 265 | 270 | 266
Participants | 90 | 73 | 78 | 68 | 155 | 154 | 171 | 145

3. Secondary Outcome: PN-Request
Description: Number of participants who were assigned to PN groups who requested patient navigation.
Time Frame: Every 10 or 30 days dependent on group randomization [up to 90 days post intervention message]
Population: Groups analyzed for this outcome are only PN groups/arms. No Patient Navigation (NoPN) groups were not analyzed for this outcome since patient navigation was not offered to those groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day
Number analyzed (Participants) | 0 | 0 | 264 | 262 | 0 | 0 | 270 | 266
Participants | 0 | 0 | 3 | 3 | 0 | 0 | 3 | 1

4. Secondary Outcome: PN-Engage
Description: Number of participants who were in PN groups who talked to a patient navigator.
Time Frame: Every 10 or 30 days dependent on group randomization [up to 90 days post intervention message]
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day
Number analyzed (Participants) | 0 | 0 | 264 | 262 | 0 | 0 | 270 | 266
Participants | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 0

5. Secondary Outcome: Opt Out
Description: Number of participants who replied to stop receiving study interventions. Participants could opt-out at any time regardless of message timing.
Time Frame: Daily [up to 90 days post intervention message]
Measure: Count of Participants; unit: Participants
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day
Number analyzed (Participants) | 261 | 264 | 264 | 262 | 265 | 265 | 270 | 266
Participants | 14 | 2 | 27 | 13 | 23 | 3 | 15 | 9

6. Secondary Outcome: Self-reported Testing
Description: Participant self-reported testing as completed. Reported only for participants who requested COVID-19 test kits from the study and responded to follow-up messages.
Time Frame: 90 days post intervention message
Population: Reported only for participants who requested COVID-19 test kits from the study and responded to follow-up messages.
Measure: Count of Participants; unit: Participants
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day
Number analyzed (Participants) | 38 | 34 | 34 | 31 | 105 | 101 | 105 | 84
Participants | 18 | 16 | 13 | 13 | 32 | 37 | 41 | 25

ADVERSE EVENTS:
Time Frame: 10 months
Description: This study was a text message based study that had little risk to participants.
Arm/Group | Conversational Agent (CA) + No Patient Navigation (NoPN) + 10 Day | Conversational Agent (CA) + No Patient Navigation (PN) + 30 Day | Conversational Agent (CA) + Patient Navigation (PN) + 10 Day | Conversational Agent (CA) + Patient Navigation (PN) + 30 Day | Text Message (TM) + No Patient Navigation (NoPN) + 10 Day | Text Message (TM) + No Patient Navigation (NoPN) + 30 Day | Text Message (TM) + Patient Navigation (PN) + 10 Day | Text Message (TM) + Patient Navigation (PN) + 30 Day
All-Cause Mortality (participants affected / at risk) | 0/261 | 0/264 | 0/264 | 0/262 | 0/265 | 0/265 | 0/270 | 0/266
Serious Adverse Events (participants affected / at risk) | 0/261 | 0/264 | 0/264 | 0/262 | 0/265 | 0/265 | 0/270 | 0/266
Other Adverse Events (participants affected / at risk) | 0/261 | 0/264 | 0/264 | 0/262 | 0/265 | 0/265 | 0/270 | 0/266

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT05533359/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT05533359/SAP_001.pdf